CLINICAL TRIAL: NCT05451355
Title: Developing a Dyadic Shared Decision Making Tool About Firearm Storage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Emily Kroshus, Research Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002944
Record Dates: First submitted 2022-06-24; First posted 2022-07-11 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Safety
Keywords: Firearms; Adolescent

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants receive a link to review an educational webpage (e.g., the AAP Firearm Storage Web Page)
  Interventions: Behavioral: AAP Firearm Storage Web Page
- Intervention Group (Experimental): Participants receive the newly developed prototype (e.g., the Family Safety Check In)
  Interventions: Behavioral: Family Safety Check-In

INTERVENTIONS:
Behavioral: Family Safety Check-In — Prototype decision aid to support within-family communication and decision making about firearm storage.
  Arms: Intervention Group
Behavioral: AAP Firearm Storage Web Page — Educational web page that discusses safe firearm storage practices.
  Arms: Control Group

SUMMARY:
Given that firearm ownership is legal, common, and valued by many people in the U.S, safe storage is important to minimize the risk of unauthorized access, injury and death. Safe storage is particularly important in households with children, as they are at elevated risk of death by unintentional injury or suicide if a gun is accessible in the home. However, only 1/3 of firearm-owning parents with children in the home report consistently safe storage. Decisions about firearm storage are complex, with perceived costs and benefits of different storage options varying by individual factors (i.e., primary reasons for firearm ownership, types of firearms), family factors (i.e., age and mental and physical health of household members), and community factors (i.e., crime and norms). Storage decisions affect all household members, and prior research finds that firearm owners who discuss storage with other family members have the safest storage practices. However, a recent survey study of firearm-owning US parents of school-aged youth (n=749) found that in only 55% of parenting dyads are both parties highly involved in the decision about how firearms are stored. In this sample, investigators observed that safe storage was more likely when both members of a parenting dyad were highly involved in the storage decision (regardless of their gender and whether one or both own firearms). However, at present firearm storage interventions are directed at individuals rather than family systems. Given the prevalence of pediatric firearm injuries and the role of within-family processes in storage safety, there is a critical need to develop a feasible, self-directed, family-centered firearm safety intervention.

The objective of the proposed short-term project is to develop and obtain preliminary data about acceptability and feasibility of a prototype of a brief decision aid for parenting dyads. The conceptual framework for the decision aid is the Ottawa Decision Support Framework, and then investigators will adapt the Ottawa Person Decision Guide for Two to this issue and for self-facilitation outside of the clinical setting.

DETAILED DESCRIPTION:
Investigators will recruit up to 400 individuals who meet the following eligibility criteria: parent or guardian of at least one child under the age of 18, lives with at least one other adult (e.g., romantic partner, parent), lives in the United States, and has at least one firearm in the home. Participants will be recruited using a Qualtrics survey panel with demographic screening questions to generate a sample of eligible individuals.

Parents will access a link to a web-based survey platform (e.g., Qualtrics) and complete a series of survey questions, they will then be randomized to view either (1) the Family Safety Check-In (intervention) or (2) the AAP Firearm Storage web page (active control). All participants will then complete the same series of additional survey questions.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian of at least one child under the age of 18
* Lives with at least one other adult (e.g., romantic partner, parent)
* Lives in the United States
* Has at least one firearm in the home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Change in communication intentions | Baseline, Immediately post-intervention
  Parent self-report of their intentions to talk with their partner about how their household stores firearms (e.g., In the next 2 weeks, do you think that you will talk with your partner about how your household stores firearms? [Response options: definitely no, probably no, probably yes, definitely yes])
Change in planning intentions | Baseline, Immediately post-intervention
  Parent self report of their intention to make a plan with theirpartner about storing firearms in their household more safely. (e.g., In the next 2 weeks, do you think that you will make a plan with your partner about storing firearms in your household more safely? By plan we mean having a discussion and deciding on something you are all expected to do. [Response options: definitely no, probably no, probably yes, definitely yes])

SECONDARY OUTCOMES:
Decision making | Baseline, Immediately post-intervention
  Self-report scales of parent how parent feels about making decisions about firearm storage (feeling informed about risks, clarity on what matters most, perceived benefits and barriers of shared decision making).

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No